CLINICAL TRIAL: NCT01988818
Title: A Mono-centre, Post CE-mark, Prospective-randomized Clinical Trial to Evaluate the Performance of a Flexible Self-adherent Absorbent Dressing Coated With a Soft Silicone Layer After Hip or Knee Arthroplasty or Primary Spine Surgery in Comparison to a Standard Wound Dressing (Cosmopor E®Steril, Fa. Hartmann)
Brief Title: Prospective, Randomized Study of 2 Different Wound Dressings
Acronym: Close
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Jan Bredow, Jan Bredow, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Köln_2013-02; University Hospital Cologne (Other: University Hospital Cologne)
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Hip-surgery; Knee-surgery; Spinal-surgery
Keywords: wound dressing; silicone; standard wound dressing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard wound dressing (Active Comparator): As comparator will be used a standard Cosmopor E®adhesive, island wound dressing (Paul Hartmann LTD)after hip or knee arthroplasty or spinal surgery
  Interventions: Device: standard wound dressing
- Mepilex® Border Post-Op (Experimental): wound dressing with Mepilex® Border Post-Op with Safetac®Technology, self-adherent soft silicone surgical dressing
  Interventions: Device: Mepilex® Border Post-Op

INTERVENTIONS:
Device: Mepilex® Border Post-Op — wound dressing with Mepilex® Border Post-Op with Safetac®Technology, self-adherent soft silicone surgical dressing
  Other Names: Mepilex® Border Post-Op with Safetac®Technology
  Arms: Mepilex® Border Post-Op
Device: standard wound dressing — standard wound dressing after hip-knee or spinal surgery
  Other Names: As comparator will be used a standard Cosmopor E®adhesive, island wound dressing (Paul Hartmann LTD)
  Arms: Standard wound dressing

SUMMARY:
The primary objective of this investigation is to evaluate the performance of a self-adhesive absorbent post-operative dressing coated with a soft silicone layer in minimize the risk of the development of blistering in subjects after hip or knee arthroplasty or spinal surgery in comparison to a standard wound dressing The secondary objectives are to evaluate:

* the performance of the dressing
* the comfort, conformability and the acceptability of the dressing
* pain before, during and after dressing removal
* the overall cost regarding dressing wear time, time to do dressing change and personal resources needed

DETAILED DESCRIPTION:
A monocentre, post CE-mark, randomized clinical trial will be conducted at the University of Cologne, Department of Orthopedics and Trauma Surgery.

Male or female subjects, 18 years and above, undergoing hip, knee or spinal surgery with an expected hospital stay for 4 days or more will be included in the trial. Individual trial duration will be for 7 days (follow-up).

Two hundred subjects will be included in the trial, i.e. 100 subjects per arm. The treatment arm (either new or standard wound dressing) will be assigned by randomization stratified by type of surgery (i.e. hip, knee or spine).

AEs/ADEs/unexpected events with the device may be documented by relevant photos at time. All photos shall include a sticker marked with subject code, visit number/date and time.

Outcome Measures

Primary variable:

• Development of blistering from day 0 to day 6 post surgery Photo documentation will be evaluated in a blinded manner by the Clinical Evaluation Committee (CEC).

Secondary variables:

* Other wound complications (i.e. leakage, inflammation, infection)
* Number of dressing changes
* Pain before, during and after dressing removal (VA scale)
* Performance and acceptability of the dressing (4 point rating scale)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18years
2. Have an expected total length of stay of 4 or more days
3. Undergoing elective primary arthroplasty of the hip or knee or spinal surgery
4. Undergoing hip surgery with a standard access
5. Give their written informed consent to participate

Exclusion Criteria:

1. Dressing size does not fit the incision area
2. Known allergy/hypersensitivity to any of the components of the dressing
3. Multi-trauma
4. Undergoing arthroplasty or spine surgery due to tumour or infection?
5. Fractures
6. Wound at the surgical site prior to surgery
7. Neurological deficit of operated side (hemiplegia, etc.)
8. Subject has documented skin disease at time of enrolment, as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Blistering | 0-6 days
  Development of blistering from day 0 to day 6 post surgery Photo documentation will be evaluated in a blinded manner by the Clinical Evaluation Committee (CEC).

SECONDARY OUTCOMES:
wound complications | 0-6 days
  Other wound complications (i.e. leakage, inflammation, infection)
dressing changes | 0-6 days
  Number of dressing changes
pain | 0-6 days
  Pain before, during and after dressing removal (VA scale)
performance and acceptability | 0-6 days
  Performance and acceptability of the dressing (4 point rating scale)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bredow, physician, Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital Cologne, Cologne, Germany

REFERENCES:
- [Derived] Bredow J, Hoffmann K, Oppermann J, Hellmich M, Eysel P, Zarghooni K. Evaluation of Absorbent Versus Conventional Wound Dressing. Dtsch Arztebl Int. 2018 Mar 30;115(13):213-219. doi: 10.3238/arztebl.2018.0213. PMID 29669676
- [Derived] Bredow J, Oppermann J, Hoffmann K, Hellmich M, Wenk B, Simons M, Eysel P, Zarghooni K. Clinical trial to evaluate the performance of a flexible self-adherent absorbent dressing coated with a soft silicone layer compared to a standard wound dressing after orthopedic or spinal surgery: study protocol for a randomized controlled trial. Trials. 2015 Mar 7;16:81. doi: 10.1186/s13063-015-0599-z. PMID 25873529